CLINICAL TRIAL: NCT01138605
Title: Continued Access to DRV/Rtv in HIV-1 Infected Children and Adolescents (Rollover Patients From C212, C228, C230)
Brief Title: TMC114-TiDP29-C232 - Study Providing Continued Access to Treatment With Darunavir (DRV)/Ritonavir (Rtv) for Children Coming From Any of the Three Ongoing Tibotec Sponsored Pediatric Studies With DRV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016768; TMC114-TiDP29-C232 (Other: Janssen Sciences Ireland UC); 2009-017013-29 (EudraCT Number); NCT02923713 (obsolete NCT alias)
Record Dates: First submitted 2010-04-08; First posted 2010-06-07 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: HIV-1 Infections
Keywords: TMC114; TMC114-TiDP29-C232; TMC114-C232; Darunavir; PREZISTA
MeSH Terms: interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (9):
- 005 (Experimental): Darunavir 400 mg tablet intake of 2 tablets once daily in combination with ritonavir
  Interventions: Drug: Darunavir
- 006 (Experimental): Ritonavir Liquid formulation 80 mg/ml taken in combination with Darunavir
  Interventions: Drug: Darunavir; Drug: Ritonavir
- 007 (Experimental): Ritonavir 100 mg capsule to be taken once or twice daily in combination with Darunavir and following the Darunavir dosing schedule
  Interventions: Drug: Darunavir; Drug: Ritonavir
- 008 (Experimental): Ritonavir 100 mg tablet to be taken once or twice daily in combination with Darunavir and following the Darunavir dosing schedule
  Interventions: Drug: Darunavir; Drug: Ritonavir
- 001 (Experimental): Darunavir Oral suspension 100 mg/ml 20 mg/kg twice daily in combination with ritonavir for body weight between 10 and 20 kg
  Interventions: Drug: Darunavir
- 002 (Experimental): Darunavir 375 mg composed via oral solution or various tablets twice daily in combination with ritonavir for body weight between 20 and 30 kg
  Interventions: Drug: Ritonavir; Drug: Darunavir
- 003 (Experimental): Darunavir 450 mg composed via oral solution or various tablets twice daily in combination with ritonavir for body weight between 30 and 40 kg
  Interventions: Drug: Ritonavir; Drug: Darunavir
- 004 (Experimental): Darunavir 600mg composed via oral solution or various tablets twice daily in combination with ritonavir for body weight as of 40 kg
  Interventions: Drug: Ritonavir; Drug: Darunavir
- 009 (Experimental): Ritonavir powder for oral suspension 10 mg/mL taken in combination with Darunavir.
  Interventions: Drug: Ritonavir

INTERVENTIONS:
Drug: Darunavir — 600mg composed via oral solution or various tablets, twice daily in combination with ritonavir, for body weight as of 40 kg
  Arms: 008
Drug: Ritonavir — Liquid formulation, 80 mg/ml, taken in combination with Darunavir
  Arms: 002
Drug: Ritonavir — 100 mg capsule, to be taken once or twice daily in combination with Darunavir and following the Darunavir dosing schedule
  Arms: 003
Drug: Darunavir — Oral suspension 100 mg/ml, 20 mg/kg twice daily in combination with ritonavir for body weight between 10 and 20 kg
  Arms: 005
Drug: Ritonavir — 100 mg tablet, to be taken once or twice daily in combination with Darunavir and following the Darunavir dosing schedule
  Arms: 004
Drug: Darunavir — 375 mg composed via oral solution or various tablets, twice daily in combination with ritonavir for body weight between 20 and 30 kg
  Arms: 006
Drug: Darunavir — 450 mg composed via oral solution or various tablets, twice daily in combination with ritonavir for body weight between 30 and 40 kg
  Arms: 007
Drug: Darunavir — 400 mg tablet, intake of 2 tablets once daily in combination with ritonavir
  Arms: 001
Drug: Ritonavir — 100 mg tablet, to be taken once or twice daily in combination with Darunavir and following the Darunavir dosing schedule
  Arms: 008
Drug: Darunavir — 375 mg composed via oral solution or various tablets, twice daily in combination with ritonavir for body weight between 20 and 30 kg
  Arms: 002
Drug: Ritonavir — Liquid formulation, 80 mg/ml, taken in combination with Darunavir
  Arms: 006
Drug: Darunavir — 450 mg composed via oral solution or various tablets, twice daily in combination with ritonavir for body weight between 30 and 40 kg
  Arms: 003
Drug: Darunavir — 600mg composed via oral solution or various tablets, twice daily in combination with ritonavir, for body weight as of 40 kg
  Arms: 004
Drug: Ritonavir — 100 mg capsule, to be taken once or twice daily in combination with Darunavir and following the Darunavir dosing schedule
  Arms: 007
Drug: Ritonavir — Ritonavir powder for oral suspension 10 mg/mL taken in combination with Darunavir.
  Arms: 009

SUMMARY:
The primary objective of this study is to continue to provide Darunavir (DRV) to pediatric patients who previously received DRV in any of three pediatric clinical studies sponsored by Tibotec Pharmaceuticals and continue to benefit from using it, in countries where DRV is not yet commercially available for the pediatric patient, is not reimbursed or cannot be accessed through another source (like access program or government program).

DETAILED DESCRIPTION:
This study has the aim to continue the provision of DRV and rtv to pediatric patients that continue to benefit from treatment with it after participation in any of three ongoing pediatric studies sponsored by Tibotec Pharmaceuticals. In addition, information on the safety of DRV and rtv in combination with other antiretroviral therapies will be assessed. At the baseline visit, inclusion and exclusion criteria will be checked to confirm eligibility. Once eligible, patients will continue treatment either on the once daily dose regimen (when coming from the TMC114-TiDP29-C230 study) or a twice daily regimen (when coming from the TMC114-C212 or TMC114-TiDP29-C228 studies). Assessments and visit frequency will take place as per local standard of care but are desirable every 3 months. The interval between two visits should not exceed 6 months. Pregnancy testing for girls having had their first menses is foreseen. In addition, it is desirable that testing includes efficacy assessments (immunology and plasma viral load) and laboratory safety assessments (hematology, biochemistry including pancreatic amylase (if available) or lipase and lipid analysis). Serious Adverse Events and certain selected Adverse Events will be collected. Treatment will be continued until one of the following criteria is met (whichever occurs first): Virologic failure, treatment limiting toxicity, loss to follow-up, withdrawal of consent or assent by the patient or withdrawal of consent by the caregiver, pregnancy, termination of the trial by the sponsor, when Darunavir becomes commercially available, is reimbursed or can be accessed through another source (as there are access program or government program) in the region the patient is living in. The sponsor advises participating centers to plan the study visits every 3 months but frequency will depend on local practice and standard of care. The sponsor has also foreseen in the study protocol a guidance on specific safety assessments to be performed as well as detailed instructions on how to deal with specific toxicities and undesirable effects. However local practice will prevail and the assessments performed may vary depending on the region the patient is participating in. Intake of study medication will happen once daily or twice daily, depending on what the patient took in the original pediatric trial. For the twice daily regimen, the regimen may be adjusted as the patient gains weight. The adult dosage regimen of 600/100 mg DRV/rtv may be administered as of 40 kg of body weight. Depending on the history of the patient, following dosages may be administered: DRV oral suspension (100mg DRV/ml), DRV tablets 75 mg, 150 mg, 600 mg, all for twice daily intake. DRV 400 mg for the once daily 800 mg intake (2 tablets per intake).DRV intake will be combined with rtv in oral suspension (80 mg rtv/ml), capsule or tablet (both 100 mg).

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed the TMC114-C212, TMC114-TiDP29-C228 or TMC114-TiDP29-C230 study and continues to benefit from DRV
* DRV is not commercially available, not reimbursed or cannot be accessed through another way
* signed informed consent by parents/caregivers or assent by the patient is available prior to inclusion

Exclusion Criteria:

* Any condition or active clinically significant disease (such as pancreas problems or cardiac problems) endangering the patient safety while being enrolled in the study
* Previously demonstrated clinically significant allergy or hypersensitivity to the study medication
* Pregnancy or breastfeeding female patients
* Specific criteria will be applicable for girls having had their first menses and for girls and boys having reached the age of sexual activity

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-10-13 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of DRV/rtv in combination with other ARVs will be summarized in terms of Mortality, all Serious Adverse Events,Adverse events leading to discontinuation and Adverse Events at least possibly related to the DRV treatment | Variable, up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (13):
- Argentina (2):
  - Buenos Aires
  - Ciudad Autonoma Buenos Aires
- Brazil (3):
  - Ribeirão Preto
  - Rio de Janeiro
  - São Paulo
- Paris, France
- Chennai, India
- South Africa (3):
  - Durban Kwazulu Natal
  - Gauteng
  - Johannesburg
- Esplugues de Llobregat, Spain
- Kyiv, Ukraine
- Birmingham, United Kingdom

REFERENCES:
- [Derived] Violari A, Masenya M, Blanche S, Vanveggel S, Hufkens V, Chetty P, Opsomer M. The DIANA Study: Continued Access to Darunavir/Ritonavir (DRV/r) and Long-Term Safety Follow-Up in HIV-1-Infected Pediatric Patients Aged 3 to < 18 Years. Drug Saf. 2021 Apr;44(4):439-446. doi: 10.1007/s40264-020-01032-0. Epub 2020 Dec 24. PMID 33367975
- See also: Continued access to darunavir/ritonavir (DRV/rtv) in HIV-1 infected children and adolescents aged 3 years and above — https://www.clinicaltrialsregister.eu/ctr-search/trial/2009-017013-29/results